CLINICAL TRIAL: NCT02120391
Title: Improving Knowledge of Medication in Ulcerative Colitis With an Iphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012 - 0726
Record Dates: First submitted 2014-04-14; First posted 2014-04-22 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Arm A) (Sham Comparator): Patients randomized to Arm A(control group) will receive an iPhone application without any of the adherence intervention turned on. The control phone application will allow patients to record their medications and how many refills they have remaining. The application will also provide patients with links about their medication.
  No adherence intervention will be done to these patients.
  Interventions: Other: iPhone Application
- Cases (Arm B) (Experimental): Patients randomized to Arm B will receive an iPhone application with the adherence intervention turned on. The study coordinator will help with the installation of the iPhone application.
  Participants in this group will not need to pay for the iPhone application.
  Interventions: Other: iPhone Application

INTERVENTIONS:
Other: iPhone Application — All subjects will receive the iPhone App on their phone however not all subjects will have the intervention (medication notifications) turned on.

SUMMARY:
The purpose of this study is to assess an iPhone application to increase adherence to maintenance medications in subjects with ulcerative colitis.

DETAILED DESCRIPTION:
Inflammatory bowel disease is a chronic condition that requires maintenance medication to maintain clinical remission. During clinical remission patient can be free of symptoms for long periods of time. Inflammatory bowel disease patients have been shown to have adherence rates around 40-60%. Non-adherence in patients in clinical remission is high with rates around 60%. Non adherence in patients in clinical remission can have significant impact because it can lead to higher rates of clinical flares and increased health care cost.

This will be a single-blinded randomized controlled trial to evaluate if patients randomized to an iPphone application vs. control can increase the adherence of their maintenance medication. The trial will last three months and we hope to enroll 99 patients.

The primary outcome will be adherence measured by the medication possession ratio. The secondary objective will be to evaluate if a validated adherence questionnaire can predict adherence in patients with inflammatory bowel disease.

Having an intervention that can increase adherence can provide better care for patients. Also having a validated survey tool can accurately identify non-adherence in inflammatory bowel disease patient would be a valuable tool for patient care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 -65 years of age.
* Diagnosed with ulcerative colitis established by history and biopsy confirmed by gastroenterology.
* On a stable dose of mesalamine for at least two months prior to entering the study
* Have an iPhone (personal iPhone)
* Patient may receive steroid or mesalamine enemas during the study only on an as needed basis

Exclusion Criteria:

• Are on more than one medication for their inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence using iPhone App | 3 months

SECONDARY OUTCOMES:
Prediction of adherence using self-administered Brief Medication Questionnaire (BMQ) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States